CLINICAL TRIAL: NCT00416260
Title: Phase 1/Phase 2, Single-Center, Controlled Study of the Effectiveness of Combined High Frequency Oscillation and Tracheal Gas Insufflation in Improving the Clinical Course of Patients With Severe Acute Respiratory Distress Syndrome
Brief Title: Combined High Frequency Oscillation and Tracheal Gas Insufflation for Severe Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Assistant Professor of Intensive Care Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10532-HFO-TGI
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Respiratory Distress Syndrome, Adult; High-Frequency Ventilation; Respiration, Artificial
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration | interventions — High-Frequency Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFO-TGI (Experimental): Patients with severe Acute Respiratory Distress Syndrome receiving sessions of high frequency oscillation and tracheal gas insufflation according to the study protocol
  Interventions: Other: High Frequency Oscillation and Tracheal Gas Insufflation
- CMV (No Intervention): Patients with severe Acute Respiratory Distress Syndrome receiving only conventional mechanical ventilation according to the study protocol

INTERVENTIONS:
Other: High Frequency Oscillation and Tracheal Gas Insufflation — Intermittent combined use of High Frequency Oscillation and Tracheal Gas Insufflation until the PaO2/inspired oxygen fraction ratio remains above than 150 mm Hg for more than 24 hours.
  Arms: HFO-TGI

SUMMARY:
In the past five years, there is a growing body of published evidence on the feasibility, and oxygenation and lung protection benefits of high frequency oscillation (HFO) in the acute respiratory distress syndrome (ARDS). The investigators have recently demonstrated the short term feasibility and additional benefits with respect to oxygenation of HFO combined with tracheal gas insufflation (TGI). In the present clinical trial, the investigators intend to test the hypothesis that HFO-TGI may result in improved respiratory physiology and clinical course compared to low tidal volume conventional mechanical ventilation in patients with severe ARDS.

DETAILED DESCRIPTION:
OBJECTIVES AND UNDERLYING HYPOTHESIS

High frequency oscillation (HFO) has beneficial physiological effects in acute respiratory distress syndrome (ARDS) [1-4]. A recent randomized controlled trial of HFO versus conventional mechanical ventilation (CMV) with traditional tidal volumes (10.1± 2.8 mL•kg-1 predicted body weight) reported a trend toward reduced 30-day mortality in the HFO arm (37% versus 52% in the CMV group; P = 0.10) [3]. To-date, HFO has not been compared to CMV with low tidal volumes (6.2 ± 1.1 mL•kg-1 predicted body weight) in ARDS [5], with respect to respiratory physiology and clinical course.

The main mechanisms of gas exchange during CMV are bulk convection and diffusion. [4, 6]. Tracheal gas insufflation (TGI) promotes CO2 elimination during CMV [7-9]. During HFO, additional gas exchange mechanisms comprise asymmetric velocity profiles, Taylor dispersion/turbulence, cardiogenic mixing, pendelluft effect, and collateral ventilation [4, 6].

We have recently shown that in patients with moderate-to-severe, primary ARDS, HFO combined with TGI (HFO-TGI) substantially improves oxygenation relative to both standard HFO and CMV according to the ARDS network protocol [5, 10]. Mean airway pressure (mPaw) was set at 1 cm H2O above the point of maximal curvature (PMC) of the expiratory pressure volume curve. During HFO-TGI, it is probably feasible to reduce mPaw, while still achieving PaO2 and peripheral oxygen saturation (SaO2) targets similar to those set by the ARDS network protocol [5]. This may result in reduced and non-traumatic ventilation pressures during HFO-TGI. Furthermore, if HFO-TGI-related gas exchange benefits are maintained during post-HFO-TGI CMV [10], then a reduction of ventilation pressures relative to the pre-HFO-TGI CMV may be feasible as well. However, the use of reduced ventilation pressures may minimize ventilator associated lung injury. In this study, we will test the hypothesis that HFO-TGI may improve the respiratory physiology and clinical course of patients with severe ARDS.

METHODS Patients

The protocol has been approved by the Scientific Committee of Evaggelismos Hospital. Informed consent will be requested from the next-of-kin of participation-eligible patients. Eligible patients should fulfill the criteria: 1) early (diagnosis established within the preceding 72 h) ARDS according to the American-European Consensus Conference Criteria [11]; 2) severe oxygenation disturbances {defined as PaO2/inspired oxygen fraction (FiO2) < 150 mm Hg}, while ventilated with a positive end-expiratory pressure (PEEP) of ≥ 8 cm H2O (criterion for severe ARDS); 3) age 18-75 years, body weight > 40 kg, and absence of a) severe air leak (i.e. > 1 chest tube per hemithorax with a persistent airleak for > 72 h); b) systolic arterial pressure of < 90 mm Hg while receiving fluids and norepinephrine at ≥ 0.5 μg/kg/min; c) significant heart disease (i.e. ejection fraction < 40 %, history of pulmonary edema, and active coronary ischemia or myocardial infarction); d) significant chronic obstructive pulmonary disease (COPD) or asthma [10]; e) intracranial abnormalities causing uncontrollable intracranial hypertension; f) chronic interstitial lung disease associated with bilateral pulmonary infiltrates; g) lung biopsy or resection on current admission; h) previous lung or bone marrow transplant, or presence of immunosuppression; i) inability to wean from prone positioning or inhaled nitric oxide; k) pregnancy or morbid obesity (i.e. body mass index > 40 kg/m2); and l) enrollment in another interventional study. Patient monitoring will include electrocardiographic lead II, hemodynamics, and SaO2. Deep sedation/neuromuscular blockade will be employed as previously described [10, 12].

CMV strategy In the 37-bed intensive care unit (ICU) of Evaggelismos hospital, a ventilatory strategy similar to the ARDS network protocol is routinely employed. Consequently, before randomization, patients will already be ventilated (Siemens 300C ventilator; or Galileo Gold, Hamilton Medical) with one of the network-protocol allowable combinations of FiO2 and PEEP [5]. Administered tidal volumes will be 5.5-7.5 mL•kg-1 predicted body weight, ventilatory rate (e.g. 20-35•min-1) will be adjusted so that pHa is kept within 7.20-7.45; the inspiration to expiration duration ratio will be 1:1 to 1:3; and the target plateau inspiratory pressure will be ≤ 30-35 cm H2O. Oxygenation goals will be PaO2 = 55-80 mm Hg or SaO2 = 88-95%.

Randomization Patients will be randomly assigned to either the CMV-group or the HFO-TGI-group. CMV-group patients will continue to receive CMV as described above. In the HFO-TGI-group, 30 min prior to HFO-TGI initiation, an inspiratory and an expiratory pressure volume curve will be consecutively constructed with the linear pressure ramp technique (whenever clinically feasible [10, 13].

HFO-TGI strategy The Sensormedics 3100B ventilator [10] will be connected to the endotracheal tube. Also, a thin Vygon TGI catheter {internal / external diameter = 1.0 / 2.0 mm, respectively [10]} will be introduced into the endotracheal tube. TGI catheter tip will be placed 0.5-1 cm beyond the endotracheal tube tip. The proximal end of the TGI catheter will be connected to an O2 flowmeter. Initial HFO settings will be as follows: 1) FiO2 = 100%, later-on titrated toward the FiO2 of preceding CMV; 2) bias flow = 30 L•min-1; 3) oscillation frequency = 4.0-5.0 Hz; 4) oscillatory pressure amplitude = arithmetical PaCO2 value during preceding CMV + 20-30 cm H2O, maximal acceptable value = 95-100 cm H2O [10]; 5) inspiratory to expiratory time ratio = 1:2; and 6) mPaw adjusted so that mean tracheal pressure = 2-3 cm H2O above the mean tracheal pressure of the preceding CMV (corresponding to an HFO mPaw of 9-10 cm H2O above the preceding CMV mPaw). Sixty to 120 secs after HFO initiation, a recruitment maneuver will be performed by pressurizing the HFO circuit at 40-45 cm H2O for 20-30 secs with oscillator piston off. HFO will then be resumed, a 3-5 cm H2O endotracheal tube cuff leak will be placed. Immediately thereafter, continuous forward thrust TGI (flow = 50% of the minute ventilation of the preceding CMV [10]) will be superimposed on the HFO.The mPaw control knob will then be adjusted to return mPaw to its originally set value. Fifteen min thereafter, arterial blood gas analysis will be performed and oscillatory pressure amplitude and oscillation frequency will be adjusted, in order to achieve a PaCO2 of < 10-15 mm Hg above the PaCO2 of the preceding CMV and to keep pHa > 7.20. After another 30-60 min, blood gas analysis will be repeated, and then, mPaw will be gradually reduced (estimated reduction rate: 0-1 cm H2O•h-1) toward a target mean tracheal pressure of up to 2-3 cm H2O lower than the mean tracheal pressure of the preceding CMV (corresponding to an HFO mPaw of 3-4 cm H2O above preceding CMV mPaw). Subsequently, TGI will be discontinued and standard HFO will be continued for 30 min. The aforementioned adjustments should permit maintenance of SaO2 = 88-95% or PaO2 = 55-80 mm Hg and of the above-described target PaCO2/pHa.

Return to CMV will be considered at the following HFO settings: mPaw adjusted so that HFO-mean tracheal pressure = up to 2-3 cm H2O lower than tracheal pressure of preceding CMV (corresponding to an HFO mPaw of 3-4 cm H2O above preceding CMV mPaw); FiO2 = FiO2 of preceding CMV; and TGI = 0 L•min-1. CMV will be resumed and continued, provided that PaO2/FiO2 is maintained at ≥ 150 mm Hg at a PEEP of ≥ 8 cm H2O. Return to HFO-TGI will be considered necessary if after 12-16 h of CMV, PaO2/FiO2 is < 150 mm Hg at a PEEP of ≥ 8 cm H2O. In the HFO-TGI-group, patients will receive repeated daily sessions of HFO-TGI until they no longer satisfy the severe ARDS criterion during CMV for > 24 h. Predicted minimum duration of HFO-TGI sessions is 6 h. For HFO-TGI-group members, total HFO-TGI duration will have to be > 12 h.

Recruitment Maneuvers:

Recruitment maneuvers (with continuous positive airway pressure of 40-50 cm H2O and a duration of 20-30 secs) will be performed as follows:

In the HFO-TGI group, recruitment maneuvers will be performed at the onset and at 3 h following the onset of each HFO-TGI session, and just prior to return to CMV. In the CMV-group, > 3 recruitment maneuvers (one every 3 h; first maneuver at 9:00 am) will be performed daily. In both groups, recruitment maneuvers will be continued as part of the early intervention period of the study protocol until resolution of severe ARDS (if achieved) or death.

Weaning from CMV:

Weaning from CMV will be by pressure-supported ventilation when a PaO2 of ≥ 60 mm Hg can be maintained at an FiO2 of ≤ 50% and a PEEP of ≤ 8 cm H2O.

Data Collection Data on demographic, physiologic, and radiographic characteristics, coexisting conditions, and medication will be recorded within 4 h prior to randomization. Physiologic, laboratory, and radiographic/imaging data will be collected daily up to 28 days post-randomization. Patients will be monitored daily for signs of failure of nonpulmonary organs and systems.

Outcome Measures are reported in the dedicated section.

In concordance with a suggestion of a recent Editorial (Intensive Care Med (2014) 40:743-745), the Original and (its revision to) the Final Form of the Study Protocol (also corresponding to NCT00637507) detailing the Pre-specified Study Planning (which explains the reason for any prior changes in the current registration data) can be found by scrolling down to the end of the following webpage: http://www.evaggelismos-hosp.gr/0010000688/%CE%B9%CF%83%CF%84%CE%BF%CF%81%CE%B9%CE%BA%CE%BF-%CE%B5%CE%B5%CF%80%CE%BD%CE%B5.html

ELIGIBILITY:
Inclusion Criteria:

* Early Acute Respiratory Distress Syndrome
* PaO2/FiO2 < 150 mm Hg at PEEP ≥ 8 cm H2O
* Age 18-75 years
* Body weight > 40 kg

Exclusion Criteria:

* More than 1 chest tube/hemithorax with persistent airleak for > 72 h)
* Systolic pressure < 90 mm Hg with fluids/norepinephrine at ≥ 0.5 μg/kg/min
* Heart disease (defined in Detailed Description)
* Chronic obstructive pulmonary disease (defined in Detailed Description)
* Intracranial abnormalities (any cause of intracranial pressure > 20 mm Hg)
* Chronic interstitial lung disease
* Lung biopsy or resection on current admission
* Previous lung or bone marrow transplant or immunosuppression
* Pregnancy or morbid obesity
* Inability to wean from prone positioning or inhaled nitric oxide
* Enrollment in another interventional study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Physiological variables (i.e. ventilation pressures and oxygenation) during the first 7-10 days following randomization | 8-10 days post-randomization
Survival to days 28 and 60 post-randomization and to Hospital Discharge | 28 days to more than 60 days post-randomization

SECONDARY OUTCOMES:
Ventilator free days | 28 days and 60 days
Number of Organ or system failure free days | 28 days and 60 days
Occurence of Barotraumas/airway injury | 28 days and 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, Lecturer, Principal Investigator — First Department of Intensive Care Medicine, University of Athens Medical School; Sotiris M Malachias, Consultant, Principal Investigator — First Department of Intensive Care Medicine, University of Athens Medical School; Charis Roussos, Professor, Study Chair — First Department of Intensive Care Medicine, University of Athens Medical School; Spyros G Zakynthinos, As Professor, Study Director — First Department of Intensive Care Medicine, University of Athens Medical School
Locations (1):
- Evaggelismos General Hospital, Athens, Attica, Greece

REFERENCES:
- [Background] Mehta S, Granton J, MacDonald RJ, Bowman D, Matte-Martyn A, Bachman T, Smith T, Stewart TE. High-frequency oscillatory ventilation in adults: the Toronto experience. Chest. 2004 Aug;126(2):518-27. doi: 10.1378/chest.126.2.518. PMID 15302739
- [Background] Ferguson ND, Chiche JD, Kacmarek RM, Hallett DC, Mehta S, Findlay GP, Granton JT, Slutsky AS, Stewart TE. Combining high-frequency oscillatory ventilation and recruitment maneuvers in adults with early acute respiratory distress syndrome: the Treatment with Oscillation and an Open Lung Strategy (TOOLS) Trial pilot study. Crit Care Med. 2005 Mar;33(3):479-86. doi: 10.1097/01.ccm.0000155785.23200.9e. PMID 15753735
- [Background] Derdak S, Mehta S, Stewart TE, Smith T, Rogers M, Buchman TG, Carlin B, Lowson S, Granton J; Multicenter Oscillatory Ventilation For Acute Respiratory Distress Syndrome Trial (MOAT) Study Investigators. High-frequency oscillatory ventilation for acute respiratory distress syndrome in adults: a randomized, controlled trial. Am J Respir Crit Care Med. 2002 Sep 15;166(6):801-8. doi: 10.1164/rccm.2108052. PMID 12231488
- [Background] Imai Y, Slutsky AS. High-frequency oscillatory ventilation and ventilator-induced lung injury. Crit Care Med. 2005 Mar;33(3 Suppl):S129-34. doi: 10.1097/01.ccm.0000156793.05936.81. PMID 15753718
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Pillow JJ. High-frequency oscillatory ventilation: mechanisms of gas exchange and lung mechanics. Crit Care Med. 2005 Mar;33(3 Suppl):S135-41. doi: 10.1097/01.ccm.0000155789.52984.b7. PMID 15753719
- [Background] Nahum A, Ravenscraft SA, Nakos G, Burke WC, Adams AB, Marcy TW, Marini JJ. Tracheal gas insufflation during pressure-control ventilation. Effect of catheter position, diameter, and flow rate. Am Rev Respir Dis. 1992 Dec;146(6):1411-8. doi: 10.1164/ajrccm/146.6.1411. PMID 1456557
- [Background] Burke WC, Nahum A, Ravenscraft SA, Nakos G, Adams AB, Marcy TW, Marini JJ. Modes of tracheal gas insufflation. Comparison of continuous and phase-specific gas injection in normal dogs. Am Rev Respir Dis. 1993 Sep;148(3):562-8. doi: 10.1164/ajrccm/148.3.562. PMID 8368624
- [Background] Nahum A, Ravenscraft SA, Nakos G, Adams AB, Burke WC, Marini JJ. Effect of catheter flow direction on CO2 removal during tracheal gas insufflation in dogs. J Appl Physiol (1985). 1993 Sep;75(3):1238-46. doi: 10.1152/jappl.1993.75.3.1238. PMID 8226536
- [Background] Mentzelopoulos SD, Roussos C, Koutsoukou A, Sourlas S, Malachias S, Lachana A, Zakynthinos SG. Acute effects of combined high-frequency oscillation and tracheal gas insufflation in severe acute respiratory distress syndrome. Crit Care Med. 2007 Jun;35(6):1500-8. doi: 10.1097/01.CCM.0000265738.80832.BE. PMID 17440419
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Murray MJ, Cowen J, DeBlock H, Erstad B, Gray AW Jr, Tescher AN, McGee WT, Prielipp RC, Susla G, Jacobi J, Nasraway SA Jr, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists, American College of Chest Physicians. Clinical practice guidelines for sustained neuromuscular blockade in the adult critically ill patient. Crit Care Med. 2002 Jan;30(1):142-56. doi: 10.1097/00003246-200201000-00021. No abstract available. PMID 11902255
- [Background] Mentzelopoulos SD, Roussos C, Zakynthinos SG. Static pressure volume curves and body posture in acute respiratory failure. Intensive Care Med. 2005 Dec;31(12):1683-92. doi: 10.1007/s00134-005-2838-3. Epub 2005 Oct 26. PMID 16249926
- [Derived] Mentzelopoulos SD, Malachias S, Zintzaras E, Kokkoris S, Zakynthinos E, Makris D, Magira E, Markaki V, Roussos C, Zakynthinos SG. Intermittent recruitment with high-frequency oscillation/tracheal gas insufflation in acute respiratory distress syndrome. Eur Respir J. 2012 Mar;39(3):635-47. doi: 10.1183/09031936.00158810. Epub 2011 Sep 1. PMID 21885390